CLINICAL TRIAL: NCT06152081
Title: A Pilot Clinical Trial Comparing the Efficacy of Caries Detection With a Novel Caries Detecting Rinse and Existing Diagnostic Tools
Brief Title: Caries Detection With Two Different Caries Detecting Devices
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00003913
Record Dates: First submitted 2023-06-13; First posted 2023-11-30 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Caries,Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- All Participants (Experimental): All participants enrolled in the study will have the two caries detecting devices used during each research visit.
  Interventions: Device: LumiCare rinse; Device: QLF Inspektor Pro Imaging

INTERVENTIONS:
Device: LumiCare rinse — The teeth being assessed will be cleaned of any debris ,plaque and calculus. The areas being assessed will be air dried. A dry field will be maintained using cotton rolls and a saliva ejector. Lumicare rinse will be applied onto the test areas for 30 seconds and the excess removed using a saliva ejector. The sites will then be rinsed with plain water for 10 seconds and excess will be removed using high volume suction. A blue curing light will then be held 1-2 inches from the test surfaces while the examiner assesses the surfaces for the presence or absence of fluorescent illumination.
Device: QLF Inspektor Pro Imaging — The teeth being assessed will be cleaned of any debris ,plaque and calculus. The areas being assessed will be air dried. A dry field will be maintained using cotton rolls and a saliva ejector. The QLF device will be positioned over the tooth surface to be tested and an image will be taken. The images will be stored automatically and assessed by the examiners for the presence of green fluorescence using the QA2 program (Version 1.25, Inspektor Research systems BV, Amsterdam, The Netherlands) . The trend in green fluorescence will also be calculated using this software algorithm.

SUMMARY:
The primary aim of this study will be to compare the effectiveness of the novel LumiCare™ rinse and with QLF in determining caries progression. The secondary aim is to compare the progression of carious lesions between patients who reported use of e-cigarettes/vapes and those who did not.

ELIGIBILITY:
Inclusion Criteria:

* Patients of TUSDM Comprehensive Care Clinic
* Adult patients over the age of 21
* Extreme/High Caries Risk classification per TUSDM Caries Management by Risk Assessment (CAMBRA) form
* Presence of 2 or more initial active primary carious lesions on a free coronal surface of any tooth by visual assessment, QLF, and LumiCare™
* Presence of at least 1 cavitated lesion
* Updated (no more than 6 months old) bite wing radiographs available.
* Patients who responded either yes/no to use of e-cigarettes/vapes
* 1 active caries, 1 inactive caries and 1 sound tooth surface.

Exclusion Criteria:

* Low or moderate caries risk classification per TUSDM CAMBRA form
* No clinically detectable carious lesions on free coronal surfaces
* No cavitated caries lesions
* Carious teeth with caries lesions concomitant with extrinsic stains, fluorosis, or developmental defects.
* Patients who responded yes to the use of conventional cigarettes or smokeless tobacco

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of two caries-detecting devices | 12 months
  Compare the effectiveness of the two caries detecting devices in their ability determining caries progression

SECONDARY OUTCOMES:
Caries progression in those who do and do not use e-cigarettes/vapes | 12 months
  Comparison of the progression of carious lesions between patients who reported use of e-cigarettes/vapes and those who did not

CONTACTS AND LOCATIONS:
Overall Officials: Karina Irusa, BDS, MS, Principal Investigator — Tufts University School of Dental Medicine
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No